CLINICAL TRIAL: NCT03092882
Title: Digital Self-Management Program for Medicare Advantage Members With Type 2 Diabetes- Impact on A1c
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Evidation Health (Industry)
Collaborators: Humana Co.Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: EH-004
Record Dates: First submitted 2017-03-22; First posted 2017-03-28 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Diabetes Self-Management Program
  Interventions: Behavioral: Diabetes Self-Management Program
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Diabetes Self-Management Program — The Diabetes Self-Management Program is a platform that includes a smart meter, access to coaching 24/7, and a mobile app and website that help members manage their diabetes. The program offers diabetes education and coaching delivered entirely through the smart meter and mobile app or website.
  Arms: Intervention

SUMMARY:
The Digital Self-Management Program for Medicare Advantage Members with Type 2 Diabetes - Impact on A1c trial is a 26-week long, prospective, intent-to-treat, 2-arm randomized controlled trial that aims to evaluate the impact of the Digital Self-Management Program on A1c levels for individuals with uncontrolled Type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Humana Medicare Advantage member
* Type 2 diabetes diagnosis
* HbA1c levels ≥ 8.0% verified by lab test

Exclusion Criteria:

* Has any of the following conditions: cancer, chronic heart failure, chronic obstructive pulmonary disease, respiratory failure, chronic kidney disease, end stage renal disease, peripheral vascular disease
* Not fluent in English
* Humana membership is part of a Full or Global risk arrangement
* Enrolled in Humana at Home Care Management

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 607 (Actual)
Dates: Start 2017-03-03 (Actual); Primary Completion 2018-02-07 (Actual); Study Completion 2018-02-07 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in A1c at 6 months | Baseline and 6 months
  Change in A1c from study baseline to study end

CONTACTS AND LOCATIONS:
Overall Officials: Jessie Juusola, PhD, Principal Investigator — Evidation Health
Locations (1):
- Evidation Health, San Mateo, California, United States

IPD SHARING:
Plan to Share IPD: No